CLINICAL TRIAL: NCT01096992
Title: A Phase I/II Clinical Trial of Fludarabine, Bendamustine, and Rituximab (FBR) in Previously Treated Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Fludarabine, Bendamustine, and Rituximab (FBR) for Relapsed Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0546; NCI-2011-01942 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Leukemia
Keywords: Chronic lymphocytic leukemia; CLL; Bendamustine; Fludarabine; Fludara; Fludarabine Phosphate; Rituximab; Rituxan
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; fludarabine; fludarabine phosphate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1 20 mg/m^2 (Experimental): Bendamustine, Fludarabine + Rituximab
  Interventions: Drug: Bendamustine; Drug: Fludarabine; Drug: Rituximab
- Phase 2 (Experimental): Bendamustine 30 mg/m^2 by vein (fixed), Days 1,2,3 + Fludarabine + Rituximab
  Interventions: Drug: Bendamustine; Drug: Fludarabine; Drug: Rituximab
- Phase 1 30 mg/m^2 (Experimental): Bendamustine, Fludarabine + Rituximab
  Interventions: Drug: Bendamustine; Drug: Fludarabine; Drug: Rituximab
- Phase 1 40 mg/m^2 (Experimental): Bendamustine, Fludarabine + Rituximab
  Interventions: Drug: Bendamustine; Drug: Fludarabine; Drug: Rituximab
- Phase 1 50 mg/m^2 (Experimental): Bendamustine, Fludarabine + Rituximab
  Interventions: Drug: Bendamustine; Drug: Fludarabine; Drug: Rituximab

INTERVENTIONS:
Drug: Bendamustine — Phase 1: Starting Dose of 20 mg/m2 IV on Days 1,2,3 (after fludarabine)
  Phase 2: 30 mg/m2 by vein (fixed) on Days 1,2,3 (after fludarabine)
  Other Names: Bendamustine HCI; Bendamustine Hydrochloride; CEP-18083; SDX-105; Treanda
Drug: Fludarabine — Course 1: 20 mg/m2 intravenous (IV) on Days 2,3,4 Courses 2-6: 20 mg/m2 IV, Days 1,2,3
  Other Names: Fludara; Fludarabine Phosphate
Drug: Rituximab — Course 1: 375 mg/m2 IV, Day 4 (after fludarabine) Courses 2-6: 500 mg/m2 IV, Day 1
  Other Names: Rituxan

SUMMARY:
The goal of Phase 1 of this clinical research study is to find the highest tolerable dose of bendamustine, combined with fludarabine and rituximab, that can be given to patients who have CLL that has been treated before.

The goal of Phase 2 of this study is to find out if this drug combination can help to control the disease. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Fludarabine and bendamustine are designed to damage the DNA (genetic material) of cancer cells, which may cause the cancer cells to die.

Rituximab is designed to attach to cancer cells and damage them, which may cause the cancer cells to die. It is also designed to cause the immune system to attack cancer cells.

Study Drug Dose Levels:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined this study. One (1) to 8 groups with 3-6 participants will be enrolled in the Phase 1 portion of the study, and up to 58 participants will be enrolled in Phase 2.

If you are enrolled in Phase 1, the dose of bendamustine you receive will depend on when you joined this study. The first group will receive the lowest dose. The next group will receive a higher dose, if the number and type of side effects was low or none. The dose of bendamustine will be increased for each new group until the highest tolerable dose is found.

If you are enrolled in Phase 2, you will receive bendamustine at the highest dose that was tolerated in Phase 1.

All participants in both phases of the study will start out with the same dose levels of fludarabine and rituximab.

If side effects occur, the study doctor may decide to lower your doses of study therapy. If you have side effects during a dose, the study staff will observe you for any other problems for 2 hours after the dose.

Study Drug Administration:

Cycles in this study are 4 weeks. All 3 study drugs are given by vein.

Cycle 1:

* On Days 1-3, bendamustine will be given over 30 minutes.
* On Days 2-4, fludarabine will be given over 30 minutes.
* On Day 4, rituximab will be given over 6-8 hours.

Cycles 2-6:

* On Day 1, rituximab will be given at a higher dose than in Cycle 1. If you tolerated the Cycle 1 dose well, your Cycles 2-6 rituximab doses may be given over 2-4 hours.
* On Days 1-3, fludarabine will be given over 30 minutes.
* On Days 1-3, bendamustine will be given over 30 minutes.

Other Drugs:

You will be given Tylenol (acetaminophen) and Benadryl (diphenhydramine hydrochloride) to take by mouth 30-60 minutes before every dose of rituximab (Cycles 1-6). These drugs are given to lower the risk of side effects.

Study Visits:

Once a week in Cycle 1 and every 2-4 weeks in Cycles 2-6, blood (about 1 tablespoon) will be drawn for routine tests.

Before Cycles 1-6, you will also have a physical exam, including measurement of your vital signs. You will be asked about any side effects you may have had.

Before Cycle 4, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a bone marrow aspiration and biopsy to check the status of the disease.
* If the doctor thinks it is needed, you will have a CT scan of the neck, chest, abdomen, and pelvis to check the status of the disease.

Length of Study Participation:

You may receive up to 6 cycles of study treatment. The study treatment will be stopped early if the disease gets worse or you experience any intolerable side effects.

End-of-Treatment Visit:

After Cycle 6 (or earlier if you stop early), the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a bone marrow aspiration and biopsy to check the status of the disease.
* If the doctor thinks the disease has completely responded, you will have a CT scan of the neck, chest, abdomen, and pelvis to confirm the response.

Follow-Up Visits:

You will have follow-up visits at the end of Month 6 and Year 1 after your last dose of study drugs, and once a year until you start a new cancer treatment. The same tests will be performed as at the end-of-treatment visit. Starting at Year 3, the follow-up tests and procedures can be done by your local doctor if that is more convenient to you.

You should tell your study doctor or staff if you start another cancer treatment after the study. If that occurs, your follow-up in this study will stop.

This is an investigational study. Both fludarabine and bendamustine are commercially available and FDA approved to treat CLL. Rituximab is commercially available and FDA approved to treat lymphoma. The use of these drugs together in this study is investigational.

Up to 82 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of CLL/Small Lymphocytic Lymphoma (SLL) and be previously treated
2. Patients must have an indication for treatment by 2008 IWCLL Criteria
3. Age >/= 16 years
4. Zubrod performance status </= 2
5. Adequate renal and hepatic function as indicated by all the following: a. serum creatinine </= 2 mg/dL AND; b. alanine aminotransferase (ALT) </= 2.5 times upper limit of normal AND; c. total bilirubin </= 2.5 times upper limit of normal
6. Patients must give written informed consent
7. Patients of childbearing potential must be willing to practice birth control during the study

Exclusion Criteria:

1. Pregnant or breast-feeding females
2. Significant co-morbidity indicated by major organ system dysfunction
3. Active, uncontrolled infection, including active hepatitis
4. Uncontrolled autoimmune hemolytic anemia (AIHA) or immune thrombocytopenia purpura (ITP)
5. Treatment including chemotherapy, chemoimmunotherapy, monoclonal antibody therapy, radiotherapy, high-dose corticosteroid therapy (Prednisone >/ 60 mg daily or equivalent), or immunotherapy within 21 days prior to enrollment or concurrent with this trial

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-04-19 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Wierda, MD, PhD, BS, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 4/2010 to 012/2013
Groups:
- Phase 1 20 mg/m^2: Bendamustine, Fludarabine + Rituximab
  Bendamustine: Phase 1: 20 mg/m^2 IV on Days 1,2,3 (after fludarabine)
  Fludarabine: Course 1: 20 mg/m^2 intravenous (IV) on Days 2,3,4 Courses 2-6: 20 mg/m^2 IV, Days 1,2,3
  Rituximab: Course 1: 375 mg/m^2 IV, Day 4 (after fludarabine) Courses 2-6: 500 mg/m^2 IV, Day 1
- Phase 1 30 mg/m^2: Bendamustine, Fludarabine + Rituximab
  Bendamustine: Phase 1: 30 mg/m^2 IV on Days 1,2,3 (after fludarabine)
  Fludarabine: Course 1: 20 mg/m^2 intravenous (IV) on Days 2,3,4 Courses 2-6: 20 mg/m^2 IV, Days 1,2,3
  Rituximab: Course 1: 375 mg/m^2 IV, Day 4 (after fludarabine) Courses 2-6: 500 mg/m^2 IV, Day 1
- Phase 1 40 mg/m^2: Bendamustine, Fludarabine + Rituximab
  Bendamustine: Phase 1: 40 mg/m^2 IV on Days 1,2,3 (after fludarabine)
  Fludarabine: Course 1: 20 mg/m^2 intravenous (IV) on Days 2,3,4 Courses 2-6: 20 mg/m^2 IV, Days 1,2,3
  Rituximab: Course 1: 375 mg/m^2 IV, Day 4 (after fludarabine) Courses 2-6: 500 mg/m^2 IV, Day 1
- Phase 1 50 mg/m^2: Bendamustine, Fludarabine + Rituximab
  Bendamustine: Phase 1: 50 mg/m^2 IV on Days 1,2,3 (after fludarabine)
  Fludarabine: Course 1: 20 mg/m^2 intravenous (IV) on Days 2,3,4 Courses 2-6: 20 mg/m^2 IV, Days 1,2,3
  Rituximab: Course 1: 375 mg/m^2 IV, Day 4 (after fludarabine) Courses 2-6: 500 mg/m^2 IV, Day 1
- Phase 2: Bendamustine 30 mg/m^2 by vein (fixed), Days 1,2,3 + Fludarabine + Rituximab
  Phase 2: 30 mg/m^2 by vein (fixed) on Days 1,2,3 (after fludarabine)
  Fludarabine: Course 1: 20 mg/m^2 intravenous (IV) on Days 2,3,4 Courses 2-6: 20 mg/m^2 IV, Days 1,2,3
  Rituximab: Course 1: 375 mg/m^2 IV, Day 4 (after fludarabine) Courses 2-6: 500 mg/m^2 IV, Day 1
Period: Overall Study
Arm/Group | Phase 1 20 mg/m^2 | Phase 1 30 mg/m^2 | Phase 1 40 mg/m^2 | Phase 1 50 mg/m^2 | Phase 2
Started | 6 | 3 | 6 | 6 | 30
Completed | 6 | 3 | 6 | 6 | 30
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 20 mg/m^2 | Phase 1 30 mg/m^2 | Phase 1 40 mg/m^2 | Phase 1 50 mg/m^2 | Phase 2 | Total
Number analyzed (Participants) | 6 | 3 | 6 | 6 | 30 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 4 | 4 | 21 | 35
  >=65 years | 2 | 1 | 2 | 2 | 9 | 16
Age, Continuous [Median (Full Range); unit: years] | 63 [46 to 82] | 64 [62 to 66] | 63 [49 to 76] | 62 [55 to 76] | 61 [46 to 73] | 62 [46 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 0 | 8 | 13
  Male | 4 | 1 | 5 | 6 | 22 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 2 | 4
  White | 5 | 3 | 6 | 5 | 27 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 3 | 6 | 6 | 30 | 51

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Bendamustine Combined With Fixed-Dose Fludarabine and Rituximab (FBR)
Description: MTD defined as highest dose level in which 6 participants have been treated with </= to 1 patient experiencing dose limiting toxicity (DLT). MTD exceeded if 2 or more of 6 patients experience grade 3 or higher, non-hematologic, non-infusion related toxicity a major organ system. DLT defined as treatment-related, grade >/= 3 non-hematologic toxicity. Hematologic toxicity grade >/= 3 that lasts longer than 42 days considered a DLT. Hematologic toxicity graded according to the 2008 IWCLL criteria for grading. Tumor lysis not considered a DLT.
Time Frame: After 4 week cycle
Population: Maximum Tolerated Dose (MTD) was not established as an objective for the phase II portion of this study and was not collected.
Measure: Number; unit: mg/m^2
Groups:
- Phase 1: Bendamustine, Fludarabine + Rituximab
  Bendamustine: Phase 1: Starting Dose of 20 mg/m2 IV on Days 1,2,3 (after fludarabine)
  Phase 2: 30 mg/m2 by vein (fixed) on Days 1,2,3 (after fludarabine)
  Fludarabine: Course 1: 20 mg/m2 intravenous (IV) on Days 2,3,4 Courses 2-6: 20 mg/m2 IV, Days 1,2,3
  Rituximab: Course 1: 375 mg/m2 IV, Day 4 (after fludarabine) Courses 2-6: 500 mg/m2 IV, Day 1
Arm/Group | Phase 1
Number analyzed (Participants) | 21
mg/m^2 | 30

2. Secondary Outcome: Overall Response Rate of Bendamustine Combined With Fixed-Dose Fludarabine and Rituximab (FBR)
Description: Overall Response is Complete response (CR) + Partial response (PR). Overall response evaluated by 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 for complete or partial response and progressive disease. Complete remission (CR), requiring absence of peripheral blood clonal lymphocytes by immunophenotyping, absence of lymphadenopathy, absence of hepatomegaly or splenomegaly, absence of constitutional symptoms and satisfactory blood counts; positive or negative minimal residual disease (MRD); Partial remission (PR), defined as ≥ 50% fall in lymphocyte count, ≥ 50% reduction in lymphadenopathy or ≥ 50% reduction in liver or spleen, together with improvement in peripheral blood counts;
Time Frame: Overall response assessed 2 months after 6th or last course if participants not able to receive all 6 intended courses of treatment.
Population: Two participants in the phase II portion of the study were not evaluable for response due to loss to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 20 mg/m^2 | Phase 1 30 mg/m^2 | Phase 1 40 mg/m^2 | Phase 1 50 mg/m^2 | Phase 2
Number analyzed (Participants) | 6 | 3 | 6 | 6 | 28
Participants | 5 | 3 | 5 | 2 | 17

ADVERSE EVENTS:
Time Frame: Adverse events captured from the time of participant consent until 30 days after the last dose of drug.
Arm/Group | Phase 1 20 mg/m^2 | Phase 1 30 mg/m^2 | Phase 1 40 mg/m^2 | Phase 1 50 mg/m^2 | Phase 2
All-Cause Mortality (participants affected / at risk) | 2/6 | 0/3 | 0/6 | 0/6 | 1/30
Serious Adverse Events (participants affected / at risk) | 4/6 | 0/3 | 4/6 | 5/6 | 16/30
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 6/6 | 6/6 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 20 mg/m^2 (N=6) | Phase 1 30 mg/m^2 (N=3) | Phase 1 40 mg/m^2 (N=6) | Phase 1 50 mg/m^2 (N=6) | Phase 2 (N=30)
Amloidosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Drug Rash (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fainting (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutropenic Fever (Infections and infestations) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 6 (7)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor Flare (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor Lysis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Acites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic Reaction Investigational Product (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated BUN (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Growth Neck (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage Bladder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural Hematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 20 mg/m^2 (N=6) | Phase 1 30 mg/m^2 (N=3) | Phase 1 40 mg/m^2 (N=6) | Phase 1 50 mg/m^2 (N=6) | Phase 2 (N=30)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 4 (4) | 3 (3) | 23 (33)
Fatigue (General disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 30 (30)
Hyperglycemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 30 (30)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 3 (3) | 2 (2) | 18 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 15 (32)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 7 (7)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 10 (17)
Edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Tumor Lysis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT01096992/Prot_SAP_000.pdf